CLINICAL TRIAL: NCT03273478
Title: pCONUS2 Treatment of Wide Neck Intracranial Aneurysms 2
Acronym: pToWin2
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Phenox GmbH (Industry)
Responsible Party: Sponsor
Other Study IDs: PTW2/PH/20170823
Record Dates: First submitted 2017-08-23; First posted 2017-09-06 (Actual); Last update posted 2018-04-05 (Actual); Status verified 2018-04

CONDITIONS: Intracranial Aneurysm
Keywords: Bifurcation aneurysm; Unruptured bifurcation aneurysm; Ruptured bifurcation aneurysm; Stent-assisted coiling; pCONUS2 Bifurcation Aneurysm Implant
MeSH Terms: conditions — Intracranial Aneurysm

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Device: Endovascular treatment of bifurcation aneurysm with pCONUS2 — Patients suffering from a bifurcation aneurysm will be treated endovascularly with the pCONUS2 device.
  * The patients do not face any additional risks by participating in the study as the treatment does not differ from the standard of care in any way.
  * The patients will only be enrolled in the study if they give their written consent.
  * If they do not wish to participate in the observational study or if they wish to withdraw from it at a later date, they will not have any disadvantages.

SUMMARY:
To assess safety and efficacy of pCONUS2 for the treatment of wide neck bifurcation aneurysms.

DETAILED DESCRIPTION:
Title: pCONUS2 Treatment of Wide Neck Intracranial Aneurysms 2

Acronym: pToWin2

Device: pCONUS2 Bifurcation Aneurysm Implant

Study design: Prospective, multicenter, single-arm clinical investigation

Purpose: To assess safety and efficacy of pCONUS2 for the treatment of wide neck bifurcation aneurysms

Duration of the study: 30 months

Sample size: 100 evaluable patients

Number of sites: max. 15

Follow-up intervals: Two independent follow-ups (after 3-6 and 7-12 months) according to site specific standard

ELIGIBILITY:
Inclusion Criteria:

1. Aneurysm status:

   * Unruptured aneurysm or
   * Ruptured aneurysm with a Hunt and Hess grade of I - III.
2. Age ≥18.
3. The patient or legal representative provides written informed consent.
4. The patient shows general compliance to follow the medical regimen and to attend follow-up examinations.
5. The target aneurysm is located at one of the following cerebral vessel bifurcations: ICA terminus, AcomA, MCA or BA.
6. Bifurcation wide neck aneurysm.
7. The dome height should allow for safe deployment of the device crown. The fundus of the aneurysm should offer enough space for the crown of the pCONUS2 to deploy.

Exclusion Criteria:

1. Vessel tortuosity precluding safe access and device deployment.
2. Stenosis within the vascular access or target vessel ≥ 50 %.
3. The target aneurysm has been previously treated with a stent or an intraaneurysmal implant beside coils.
4. The treatment plan for the target aneurysm includes the use of additional intra- and/or extraaneurysmal temporary or permanent implants other than coils.
5. More than one intracerebral aneurysm requires the treatment within the following 6 months.
6. Imaging evidence of an arteriovenous cerebrovascular malformation or a dural fistula.
7. Any physical, medical or psychiatric condition of the patient interfering with the adherence of the requirements and follow-up regimen of the study.
8. Any neurological disorder with progressive neurological symptoms, except attributable to a compressive effect of the target aneurysm.
9. Current involvement in another study or trial.
10. Women of child bearing potential or breast-feeding who cannot provide a negative pregnancy test.
11. Known allergy to the components of device, study medication or contrast media that cannot be controlled medically.
12. A medical condition interfering with a dual antiplatelet treatment.
13. Known coagulopathy.
14. Intracranial hemorrhage in the past 30 days apart from the target aneurysm.
15. Ischemic stroke in the past 30 days.
16. Myocardial infarction in the past 30 days.
17. Major surgery in the past 30 days.
18. Evidence of active infection at time of treatment.
19. Co -morbidities or conditions with a life expectancy less than 12 months.
20. Additional Exclusion criteria for ruptured aneurysm at the acute phase:

    1. The patient is clinically severely affected (Hunt and Hess grade IV and V).
    2. Severe vasospasm is proven during angiography.
    3. Proven parenchymal hemorrhage by CT or MRI.
    4. Proven subdural hematoma by CT or MRI.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients harbouring an unruptured or ruptured bifurcation aneurysm, in which pCONUS2-assisted coiling was judged to be the most appropriate treatment
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2018-12 (Estimated); Primary Completion 2020-12 (Estimated); Study Completion 2021-12 (Estimated)

PRIMARY OUTCOMES:
Effectiveness: Aneurysm occlusion (complete or neck remnant) | Change from post-procedure to 12 months
  Assessment by Raymond-Roy occlusion scale
Safety: Major stroke (ischemic or hemorrhagic) or neurological death related to the treatment of the target aneurysm | within 12 months

SECONDARY OUTCOMES:
Effectiveness: The "Effectiveness endpoint" is assessed throughout the intervention and is assessed as "number/amount of": | at the time of the procedure
  - To place pCONUS2 in the desired location
Effectiveness: The "Effectiveness endpoint" is assessed throughout the intervention and is assessed as "number/amount of": | at the time of the procedure
  - Correct opening of the device (crown and shaft)
Effectiveness: The "Effectiveness endpoint" is assessed throughout the intervention and is assessed as "number/amount of": | at the time of the procedure
  - To perform aneurysm occlusion without obliteration of side branches
Effectiveness: The "Effectiveness endpoint" is assessed throughout the intervention and is assessed as "number/amount of": | at the time of the procedure
  - To detach the device at the end of the procedure
Safety Intra-Procedural Complications The "Safety Intra-Procedural Complications" endpoint is assessed throughout the intervention and is assessed as "number/amount of": | at the time of the procedure
  - Vessel perforation
Safety Intra-Procedural Complications The "Safety Intra-Procedural Complications" endpoint is assessed throughout the intervention and is assessed as "number/amount of": | at the time of the procedure
  - Target aneurysm perforation with microcatheter or guidewire
Safety Intra-Procedural Complications The "Safety Intra-Procedural Complications" endpoint is assessed throughout the intervention and is assessed as "number/amount of": | at the time of the procedure
  - Target aneurysm perforation with pCONUS2
Safety Intra-Procedural Complications The "Safety Intra-Procedural Complications" endpoint is assessed throughout the intervention and is assessed as "number/amount of": | at the time of the procedure
  - Target aneurysm perforation with coils
Safety Intra-Procedural Complications The "Safety Intra-Procedural Complications" endpoint is assessed throughout the intervention and is assessed as "number/amount of": | at the time of the procedure
  - Thromboembolism
Safety Intra-Procedural Complications The "Safety Intra-Procedural Complications" endpoint is assessed throughout the intervention and is assessed as "number/amount of": | at the time of the procedure
  - Dissection of any access vessel
Safety Post-Procedural Complications The "Safety Post-Procedural Complications" endpoint is assessed throughout the intervention and is assessed as "number/amount of": | Change 1day post procedure up to 12months
  - Frequency of new parenchymal hemorrhage
Safety Post-Procedural Complications The "Safety Post-Procedural Complications" endpoint is assessed throughout the intervention and is assessed as "number/amount of": | Change 1day post procedure up to 12months
  - Frequency of new subarachnoid hemorrhage
Safety Post-Procedural Complications The "Safety Post-Procedural Complications" endpoint is assessed throughout the intervention and is assessed as "number/amount of": | Change 1day post procedure up to 12months
  - Frequency of new ischemic stroke
Safety Post-Procedural Complications The "Safety Post-Procedural Complications" endpoint is assessed throughout the intervention and is assessed as "number/amount of": | Change 1day post procedure up to 12months
  - Rupture of the target aneurysm
Safety Post-Procedural Complications The "Safety Post-Procedural Complications" endpoint is assessed throughout the intervention and is assessed as "number/amount of": | Change 1day post procedure up to 12months
  - Rate of in-stent-stenosis
Safety Post-Procedural Complications The "Safety Post-Procedural Complications" endpoint is assessed throughout the intervention and is assessed as "number/amount of": | Change 1day post procedure up to 12months
  - Rate of in-stent-thrombosis